CLINICAL TRIAL: NCT02289326
Title: Biomarker Monitoring for a Young Individual Carrying a TP53 Gene Mutation in a Familial High-Cancer Predisposition Setting
Brief Title: Biomarker Monitoring in TP53 Mutation Carriers
Status: Completed | Type: Observational
Sponsor: Scripps Health (Other)
Collaborators: J. Craig Venter Institute (Other)
Responsible Party: Principal Investigator, Laura Goetz, Staff Surgeon, Scripps Health
Other Study IDs: Scripps IRB 14-6419
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Li-Fraumeni Syndrome; Hereditary Cancer Syndromes; TP53 Gene Germline Mutation Carrier
MeSH Terms: conditions — Li-Fraumeni Syndrome; Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * DNA and RNA from blood
  * Stool samples for microbiome analysis
  * Urine samples for microbiome and general biomarker analysis
  * Saliva samples for microbiome and general biomarker analysis
  * Blood for general biomarker and metabolite profiling
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Purpose

This study is an 'N-of-one' observational study focusing on individuals with a hereditary predisposition to cancer due to a genetic mutation in the TP53 gene. An individual with this mutation has a >90% chance of developing many different forms of cancer in their lifetime. Since germline TP53 gene mutation carriers are highly susceptible to cancer, cancer prevention strategies and early cancer detection strategies are crucial. Unfortunately, the current standard of care for monitoring germline TP53 gene mutation carriers for early signs of cancer is yearly MRI scans and intermittent blood draws. Villani et al. showed that standard monitoring is inadequate and introduced a more sophisticated protocol for early cancer detection. We extended the Villani et al. protocol to include a number of markers for early detection and are currently vetting their utility, in terms of their inherent variability, patient tolerability of frequent interrogation, and ability to show changes that might indicate a need for further examination.

In addition to the markers being collected, important covariate information, such as diet, sleep, and activities are being collected (via, e.g., wearable wireless devices) in order to take them into account in assessing the levels of the markers at a single data collection time or over time. One important aspect of the protocol is to identify changes, rather than specific levels, in marker status over time for an individual that might be indicative of tumor formation, essentially exploiting the concept of 'personalized thresholds' discussed by Drescher et al.

If any indication of the presence of a cancer, tumorigenic process, or general sign of ill-health is observed, the protocol calls for a discussion of the findings among the research team, followed by a discussion between the clinical lead on the research team and the primary care provider and/or specialists overseeing a participating patient's care, possible validation of the assay(s) motivating the discussions, and a decision on how to intervene on the part of the primary care provider and/or specialists.

DETAILED DESCRIPTION:
Individuals who carry certain germline TP53 gene mutations are highly susceptible to cancer and are likely to develop any one, or many, cancer types during their lifetimes. Prevention strategies and early tumor detection strategies are crucial for such individuals. It has been shown by Villani et al. that aggressive monitoring of markers of cancer can lead to much better outcomes (e.g., earlier detection of cancer) than standard monitoring protocols. However, the choice of markers for use in early detection that can indicate the presence of cancer and surveillance and monitoring strategies of patients or individuals with specific cancer predispositions, such as inherited cancer syndromes, is complex. This choice is often guided by the observed utility of a set of markers among a broader list of potential markers in large-scale population-level clinical studies. However, the utility of an early detection or surveillance strategy based on a set of markers in the population at large does not necessarily translate to the utility of those markers for a particular individual. This phenomenon is even more problematic for individuals with rare hereditary cancer syndromes and conditions, such as individuals with germline TP53 gene mutations, as these individuals are highly susceptible to different types of cancer over their lifetimes. Even among individuals with TP53 mutations there is variation in the age-of-onset of cancers due to other factors, such as exposures to carcinogenic substances and the presences of other susceptibility mutations (Arrifin et al. 2015). In addition, given that individuals with inherited TP53 mutations are indeed rare, there are no large-scale studies that have been pursued to identify sets of markers that might be useful for monitoring TP53 mutation carriers going forward for signs of cancer and or disease generally.

Specifically, individuals who inherit DNA sequence variants in the TP53 gene have a greater than 90% chance of developing cancers in their lifetimes and often develop multiple sequential cancers during their lives. Women who carry a TP53 mutation have an 82% chance of developing cancer before age 45 (Chompret A et al. 2000) and, in general, the average age of onset of cancer for individuals carrying TP53 mutations is 28 years old, but these statistics do not take into account other factors, such as the type of mutation present and the genetic background and settings in which the carriers live. (Ruijs et al. 2010; Sagne et al. 2014; Petitjean et al. 2007) Individuals who ultimately develop cancer and harbor inherited TP53 gene mutations are described in the medical literature as having 'Li-Fraumeni Syndrome'. Unfortunately, TP53 mutation-carrying relatives of individuals with either frank Li-Fraumeni syndrome or who carry mutations in the TP53 gene (that have not yet developed cancer) have an even more elevated risk of developing cancer.(Hwang et al. 2003; Nichols et al. 2001) In addition, it has been shown that 'anticipation' occurs in families with Li-Fraumeni syndrome, such that the age of onset of cancer formation is earlier from generation to generation, putting those TP53 mutation carriers with older relatives who developed early onset cancer at even greater risk of developing cancer early in life. (Trkova et al. 2002; Arrifini et al. 2015)

In light of these findings, individual carriers of TP53 mutations with siblings who have developed Li-Fraumeni syndrome, and who are in families in which individuals in older generations have had early onset cancer, are much more likely to develop very early onset cancers and should be monitored closely for signs of cancer. In fact, the documented age-of-onset of specific cancers has been described in the literature. Table 1 shows the ranges of the average age-of-onset of different cancers depending on the measured activation levels of the mutant TP53 protein, based on the data described in the study by Petitjean et al. (2007) Note first that most TP53 mutation carriers develop multiple cancers over their lifetimes, such that the age-of-onsets of the cancers in Table 1 may be associated with a second or third cancer developed by a carrier. Second, note that categories such as 'soft tissue sarcoma' refer to a number of types of cancer and not a single cancer. These facts suggest that monitoring such individuals for early signs of cancer, even before adulthood, should be of benefit, especially for soft tissue, brain, and bone sarcomas. Importantly, it has been shown that early detection of cancers in carriers of TP53 mutations, or those with frank Li-Fraumeni syndrome, can dramatically enhance survival and the effectiveness of therapeutic interventions, as described by Villani et al. (2011) among others. However, sophisticated and comprehensive patient monitoring schemes that can facilitate the detection of early signs of cancer in individuals carrying TP53 mutations are lacking, although the few markers used in the study by Villani et al. (2011) were shown to have promise. In addition, the currently accepted and insurance-reimbursable monitoring practices for TP53 mutation carriers is one whole body image per year, which is simply inadequate and has in fact been shown to be inadequate in the clinical study by Villani et al. (2011)

As a result of these facts, the current project was designed to develop a prototype longitudinal 'biomarker' (e.g., blood based proteins) and 'biometric' (e.g., imaging or wearable wireless device) monitoring strategy for carriers of the TP53 mutation with an even more pronounced predisposition to cancer due to familial aggregation of cancer. This monitoring strategy could be useful in identifying changes in those biomarkers that might either reflect cancer formation or health-related phenomena that may exacerbate susceptibility to cancer. The project will leverage different markers, assays and devices, as well the development of an analysis and prototype visualization method for drawing inferences from the marker and device data. Ultimately, the protocol will be focused on the objective, statistical evidence-based assessment of the utility of biomarker-based surveillance methods for an individual subject carrying a TP53 mutation in a high-cancer susceptibility setting (e.g., a sibling with Li-Fraumeni syndrome and familial cancers in older generations). The protocol will include the vetted markers described by Villani et al.(1) as well as a more comprehensive set of markers, biometrics and procedures in order to increase the likelihood of detecting values or changes in the status of these markers of likely biomedical importance. Since over 50% (4/7) of the cancer survivors successfully monitored in the Villani et al. (2011) study were under age 20, the fact that the age-of-onset of cancer among TP53 mutation carriers is lowest for those with a family history of Li-Fraumeni and early onset cancers, and the published reports state age-of-onset of cancer among TP53 mutation carriers is so low (e.g., Table 1), we believe that deploying this protocol in minors and children is justified. Since many of the biomarkers to be studied are likely to have a genetic basis, it makes sense to collect phenotypes and biosamples from family members of the target patient so that their values can act as control values for the target patient's values.

The markers and frequency with which they are being collected via the protocol for the currently enrolled patient include:

* Whole body Magnetic Resonance Imaging (MRI) analyses every 4-6 months
* Focused bilateral breast MRI every 6 months
* Abdominal ultrasound imaging every 6 months
* Stool microbiome via shotgun sequencing every two weeks
* Extensive blood metabolite profiling once a month
* Circulating cell-free DNA once a month
* DNA repair assay results from blood cells once a month
* Literature-backed early cancer detection blood-based markers once every two months (17-OH-pregnenolone, testosterone, progesterone, 11 deoxycortisol, deoxycorticosterone (DOC), beta-2-microglobulin, carcinoembryonic antigen (CEA), Cancer Antigen 125 (CA-125), β-human chorionic gonadotropin(β-HCG), alpha-fetoprotein, 17-OH-progesterone, androstenedione, dehydroepiandrosterone (DHEA), lactate dehydrogenase).
* Complete blood count information once every two months
* Serum electrolyte and liver function tests once every two months (sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatinine, glucose, calcium, albumin, total protein, bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase)

This proposed, single-subject, or 'N-of-1' study design will involve longitudinal data collections (i.e., repeated samplings) on the TP53 carrier to detect likely health-informative changes over time. We emphasize that many of the biomarkers and biometrics to be studied have the potential to detect cancer, but may also simply provide indications of health status changes generally and as such we envision the proposed study as one focusing on the prototyping and implementation of a system for monitoring biomarkers that may detect tumor formation or indicate health status changes that could warrant further scrutiny.

Table 1.

Colorectal 36.3 - 52years Breast 33.3 - 42.7years Soft Tissue Sarcoma 17.3 - 20.6years Brain Tumor 23.6 - 26.2years Ostosarcoma 16.9 - 17.7years Adrenocortical 3.2 - 4.6years Lung 46.1 - 48.8years

ELIGIBILITY:
Inclusion Criteria:

1. Any individual and their family with a known functionally significant germline TP53 mutation susceptible to Li-Fraumeni Syndrome.
2. Any individual and their family with a known hereditary cancer syndrome.

Exclusion Criteria:

1. No functionally significant germline TP53 gene mutation.
2. Inability to tolerate intensive biomonitoring.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with functionally significant germline TP53 gene mutations who are susceptible to Li-Fraumeni Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Development of cancer | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Schork, PhD, Principal Investigator — J. Craig Venter Institute; Victoria Magnuson, PhD, Study Director — J. Craig Venter Institute
Locations (1):
- Scripps Clinic Medical Group, La Jolla, California, United States

REFERENCES:
- [Background] Villani A, Tabori U, Schiffman J, Shlien A, Beyene J, Druker H, Novokmet A, Finlay J, Malkin D. Biochemical and imaging surveillance in germline TP53 mutation carriers with Li-Fraumeni syndrome: a prospective observational study. Lancet Oncol. 2011 Jun;12(6):559-67. doi: 10.1016/S1470-2045(11)70119-X. Epub 2011 May 19. PMID 21601526
- [Background] Chompret A, Brugieres L, Ronsin M, Gardes M, Dessarps-Freichey F, Abel A, Hua D, Ligot L, Dondon MG, Bressac-de Paillerets B, Frebourg T, Lemerle J, Bonaiti-Pellie C, Feunteun J. P53 germline mutations in childhood cancers and cancer risk for carrier individuals. Br J Cancer. 2000 Jun;82(12):1932-7. doi: 10.1054/bjoc.2000.1167. PMID 10864200
- [Background] Ruijs MW, Verhoef S, Rookus MA, Pruntel R, van der Hout AH, Hogervorst FB, Kluijt I, Sijmons RH, Aalfs CM, Wagner A, Ausems MG, Hoogerbrugge N, van Asperen CJ, Gomez Garcia EB, Meijers-Heijboer H, Ten Kate LP, Menko FH, van 't Veer LJ. TP53 germline mutation testing in 180 families suspected of Li-Fraumeni syndrome: mutation detection rate and relative frequency of cancers in different familial phenotypes. J Med Genet. 2010 Jun;47(6):421-8. doi: 10.1136/jmg.2009.073429. PMID 20522432
- [Background] Sagne C, Marcel V, Bota M, Martel-Planche G, Nobrega A, Palmero EI, Perriaud L, Boniol M, Vagner S, Cox DG, Chan CS, Mergny JL, Olivier M, Ashton-Prolla P, Hall J, Hainaut P, Achatz MI. Age at cancer onset in germline TP53 mutation carriers: association with polymorphisms in predicted G-quadruplex structures. Carcinogenesis. 2014 Apr;35(4):807-15. doi: 10.1093/carcin/bgt381. Epub 2013 Dec 11. PMID 24336192
- [Background] Petitjean A, Achatz MI, Borresen-Dale AL, Hainaut P, Olivier M. TP53 mutations in human cancers: functional selection and impact on cancer prognosis and outcomes. Oncogene. 2007 Apr 2;26(15):2157-65. doi: 10.1038/sj.onc.1210302. PMID 17401424
- [Background] Hwang SJ, Lozano G, Amos CI, Strong LC. Germline p53 mutations in a cohort with childhood sarcoma: sex differences in cancer risk. Am J Hum Genet. 2003 Apr;72(4):975-83. doi: 10.1086/374567. Epub 2003 Feb 27. PMID 12610779
- [Background] Nichols KE, Malkin D, Garber JE, Fraumeni JF Jr, Li FP. Germ-line p53 mutations predispose to a wide spectrum of early-onset cancers. Cancer Epidemiol Biomarkers Prev. 2001 Feb;10(2):83-7. PMID 11219776
- [Background] Trkova M, Hladikova M, Kasal P, Goetz P, Sedlacek Z. Is there anticipation in the age at onset of cancer in families with Li-Fraumeni syndrome? J Hum Genet. 2002;47(8):381-6. doi: 10.1007/s100380200055. PMID 12181637
- [Background] McBride KA, Ballinger ML, Killick E, Kirk J, Tattersall MH, Eeles RA, Thomas DM, Mitchell G. Li-Fraumeni syndrome: cancer risk assessment and clinical management. Nat Rev Clin Oncol. 2014 May;11(5):260-71. doi: 10.1038/nrclinonc.2014.41. Epub 2014 Mar 18. PMID 24642672
- [Background] Drescher CW, Shah C, Thorpe J, O'Briant K, Anderson GL, Berg CD, Urban N, McIntosh MW. Longitudinal screening algorithm that incorporates change over time in CA125 levels identifies ovarian cancer earlier than a single-threshold rule. J Clin Oncol. 2013 Jan 20;31(3):387-92. doi: 10.1200/JCO.2012.43.6691. Epub 2012 Dec 17. PMID 23248253
- [Background] Ariffin H, Hainaut P, Puzio-Kuter A, Choong SS, Chan AS, Tolkunov D, Rajagopal G, Kang W, Lim LL, Krishnan S, Chen KS, Achatz MI, Karsa M, Shamsani J, Levine AJ, Chan CS. Whole-genome sequencing analysis of phenotypic heterogeneity and anticipation in Li-Fraumeni cancer predisposition syndrome. Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15497-501. doi: 10.1073/pnas.1417322111. Epub 2014 Oct 13. PMID 25313051